CLINICAL TRIAL: NCT03588078
Title: A Phase 1b/2 Study to Evaluate the Safety and Efficacy of APR-246 in Combination With Azacitidine for the Treatment of Mutation TP53 (TP53) Mutant Myeloid Neoplasms
Brief Title: Study of the Safety and Efficacy of APR-246 in Combination With Azacitidine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-APR246
Record Dates: First submitted 2018-06-20; First posted 2018-07-17 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Myelodysplastic Syndrome With Gene Mutation; Acute Myeloid Leukemia With Gene Mutations; Myeloproliferative Neoplasm; Chronic Myelomonocytic Leukemia
Keywords: Azacitidine
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic | interventions — eprenetapopt; Azacitidine

STUDY DESIGN:
Intervention Model Description: Participants will receive one dose of protocol therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- combination of APR246 and azacitidine (Experimental): Following completion of the Dose Finding Phase, we will conduct a dose expansion, whereby patients will be treated with APR-246 administered at the maximum tolerated dose (MTD) with azacitidine on a 28 day cycle utilizing the same dosing as in Phase 1b
  Interventions: Drug: APR-246; Drug: Azacitidine

INTERVENTIONS:
Drug: APR-246 — Azacitidine at maximum tolerated dose. APR246 at the Dose limited Toxicity (DLT) dose
  Other Names: PRIMA-1MET; Methylated analogue to PRIMA-1
Drug: Azacitidine — azacitidine is administered subcutaneously (SC) or via IV at 75 mg/m2
  Other Names: Mylosar; Vidaza

SUMMARY:
The main purpose of this study is to determine the safe and efficacy of APR-246 in combination with azacitidine as well as to see complete remission of this patients

DETAILED DESCRIPTION:
Patients will be treated for a total of 6 cycles.For patients responding or who have stable disease following cycle 6, treatment may continue until one of the following criteria applies:

* Inter-current illness that prevent further administration of treatment
* Unacceptable adverse event(s)
* Participant decides to withdraw from the study,
* general or specific changes in the participant's condition render the participant unacceptable for further treatment in the judgment of the investigator.
* Evidence of disease progression by international working Group (IWG) 2006 criteria.
* participants who wish not to continue treatment at time of disease assessment at end of cycle 6 will complete their end of treatment visit upon completion of cycle 6

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the Informed Consent (ICF) and is able to comply with protocol requirements.
2. Patient has adequate organ function as defined by the following laboratory values:

   1. Serum creatinine ≤ 2 x upper limit of normal (ULN)
   2. Total serum bilirubin < 1.5 x ULN or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert's Syndrome or hemolysis or who required regular blood transfusions
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN
3. Age ≥18 years at the time of signing the informed consent form
4. Documented diagnosis of myelodysplastic syndrome (MDS), MDS/ myeloproliferative neoplasm (MPN), chronic myelomonocytic leukemia (CMML) by World Health organization (WHO) criteria or non-proliferative AML (ie with WBC < 20 G/l)
5. Documentation of a TP53 gene mutation by next-generation sequencing (NGS) based on central or local evaluation.
6. Revised International Prognostic Scoring System (IPSS-R) criteria for Intermediate, High-risk or Very High-risk.
7. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 is required.
8. If of childbearing potential, negative pre-treatment urine or serum pregnancy test.
9. If of childbearing potential (males and females), willing to use an effective form of contraception such as latex condom, hormonal birth control, intrauterine device or double barrier method during chemotherapy treatment and for at least six months thereafter.

Exclusion Criteria:

1. Patient has a known history of HIV or active hepatitis B or active hepatitis C infection (testing not mandatory).
2. Patient has any of the following cardiac abnormalities (as determined by treating MD):

   1. symptomatic congestive heart failure
   2. myocardial infarction ≤ 6 months prior to enrollment
   3. unstable angina pectoris
   4. serious uncontrolled cardiac arrhythmia
   5. QTc ≥ 470 msec (≥ 500 msec in the presence of RBBB) calculated from a mean of 3 ECG readings using Fridericia's correction (QTcF = QT/RR0.33)
   6. bradycardia (<40 bpm)
   7. known left ventricular ejection fraction (LVEF) < the institution lower limit of normal as assessed by ECHO
   8. clinically significant pericardial disease
   9. electrocardiographic evidence of acute ischemia
   10. familial history of long QT syndrome
3. Concomitant malignancies or previous malignancies with less than a 1-year disease free interval at the time of signing consent. Patients with adequately resected basal or squamous cell carcinoma of the skin, or adequately resected carcinoma in situ (e.g. cervix) may enroll irrespective of the time of diagnosis.
4. Prior exposure to azacitidine, decitabine or investigational hypomethylating agent
5. Use of cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of MDS, MDS/MPN, CMML or AML within 14 days of the first day of study drug treatment.
6. No concurrent use of erythroid stimulating agents, Granulocyte-colony stimulating Factor (G-CSF), Granulocyte Macrophage-colony stimulating factor (GM-CSF) is allowed during study except in cases of febrile neutropenia where G-CSF can be used for short term. Growth factors must be stopped 14 days prior to study.
7. Patients with history of allogeneic stem cell transplantation.
8. Pregnant women are excluded from this study because APR-246 has not been studied in pregnant subjects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with APR-246, breastfeeding should be discontinued if the mother is treated with APR-246.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 8 months
  overall survival at complete remission

SECONDARY OUTCOMES:
Duration of response | minimum 24 months it is defined as the time between achieving response and progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fenaux, Principal Investigator — service Hématologie Séniors Hôpital Saint Louis
Locations (7):
- France (7):
  - Bruno Quesnel, Lille
  - Dr Pierre Peterlin and Pr Patrice Chevalier, Nantes
  - Hôpital Archet 1, Nice
  - Hôpital Saint Louis - Hématologie Séniors, Paris
  - Hôpital Cochin/Service d'Hématologie, Paris
  - Aspasia Stamatoullas, Rouen
  - Odile Beyne Rosy, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cluzeau T, Sebert M, Rahme R, Cuzzubbo S, Lehmann-Che J, Madelaine I, Peterlin P, Beve B, Attalah H, Chermat F, Miekoutima E, Rauzy OB, Recher C, Stamatoullas A, Willems L, Raffoux E, Berthon C, Quesnel B, Loschi M, Carpentier AF, Sallman DA, Komrokji R, Walter-Petrich A, Chevret S, Ades L, Fenaux P. Eprenetapopt Plus Azacitidine in TP53-Mutated Myelodysplastic Syndromes and Acute Myeloid Leukemia: A Phase II Study by the Groupe Francophone des Myelodysplasies (GFM). J Clin Oncol. 2021 May 10;39(14):1575-1583. doi: 10.1200/JCO.20.02342. Epub 2021 Feb 18. PMID 33600210